CLINICAL TRIAL: NCT00228254
Title: Vitamin A and Zinc: Prevention of Pneumonia (VAZPOP) Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Corporacion Ecuatoriana de Biotecnologia (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: R01HD038327-01 (NIH); R01HD038327 (NIH)
Record Dates: First submitted 2005-09-23; First posted 2005-09-28 (Estimated); Last update posted 2005-09-28 (Estimated); Status verified 2005-09

CONDITIONS: Pneumonia; Diarrhea; Acute Upper Respiratory Tract Infections
Keywords: acute respiratory infection; acute lower respiratory infection; diarrhea
MeSH Terms: conditions — Pneumonia; Diarrhea | interventions — Zinc; Vitamin A

INTERVENTIONS:
Drug: Zinc (12.5 mg/day)
Drug: vitamin A 10,000 IU per week

SUMMARY:
Children with malnutrition are often low in some nutrients, like zinc or vitamin A, that could help them fight off infections like pneumonia. Our study was designed to see if children who got supplements of zinc or vitamin A had fewer infections.

DETAILED DESCRIPTION:
The Vitamin A and Zinc: Prevention of Pneumonia (VAZPOP) study was a multi-year nutritionally-stratified, placebo-controlled, double-blind study of low-dose vitamin A and/or zinc in 2,582 normal and malnourished urban children aged 6 to 36 months in Quito, Ecuador. Four group of ~ 645 children were enrolled in 2000, 2001, 2002, and 2003 with each child participating for up to 50 weeks. Children were visited 4 days each week. Outcome measures were pneumonia, other respiratory tract infections, diarrheal disease, and growth.

ELIGIBILITY:
Inclusion Criteria:

Age 6 to 36 months at the time of enrollment No recent vitamin or micronutrient use Residence of 1 year or longer in the neighborhood Full and free written consent No clinical evidence of zinc or vitamin A deficiency Absence of severe malnutrition such as weight < or = to 60% of expected weight

-

Exclusion Criteria:

Age less than 6 months or greater than 36 months at enrollment Recent vitamin or micronutrient use Residence for less than 1 year in neighborhood Lack of full and free consent Any evidence of zinc or vitamin A deficiency Severe malnutrition

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2582
Dates: Start 2000-01; Study Completion 2004-06

PRIMARY OUTCOMES:
Incidence of acute lower respiratory infection (pneumonia)
Growth

SECONDARY OUTCOMES:
Additive or synergistic effects of zinc and vitamin A
Incidence of diarrheal disease
Incidence of other respiratory infections

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey K Griffiths, MD MPH&TM, Principal Investigator — Tufts University School of Medicine
Locations (2):
- Tufts University School of Medicine, Boston, Massachusetts, United States
- Corporacion Ecuatoriana de Biotecnologia, Quito, Pinchincha, Ecuador

REFERENCES:
- [Derived] Imdad A, Rogner J, Sherwani RN, Sidhu J, Regan A, Haykal MR, Tsistinas O, Smith A, Chan XHS, Mayo-Wilson E, Bhutta ZA. Zinc supplementation for preventing mortality, morbidity, and growth failure in children aged 6 months to 12 years. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD009384. doi: 10.1002/14651858.CD009384.pub3. PMID 36994923